CLINICAL TRIAL: NCT06523296
Title: Study of the Relationship Between the Presence of Anti-AChR Antibodies in the Cerebrospinal Fluid and the Presence of Neurocognitive Disorder in Myasthenic and Alzheimers's Patients.
Brief Title: Presence of Anti-RACH Antibodies and Neurocognitive Disorder in Myasthenic or Alzheimers's Patients.
Acronym: ARN-MA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-AOI-08
Record Dates: First submitted 2024-07-23; First posted 2024-07-26 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease; Myasthenia
Keywords: Anti-RACH antibodies; Myasthenia; Alzheimer's Disease; neurocognitve disorder
MeSH Terms: conditions — Alzheimer Disease | interventions — Amyloid beta-Protein Precursor

STUDY DESIGN:
Intervention Model Description: MYASTHENIA, ALZHEIMER'S DISEASES, healthy control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adults with Alzheimer's disease (Experimental)
  Interventions: Procedure: Adults with Alzheimer's disease
- Adults with Myasthenia (Experimental)
  Interventions: Procedure: Adults with Myasthenia
- healthy volonteer (Experimental)
  Interventions: Other: Healhty controls

INTERVENTIONS:
Procedure: Adults with Alzheimer's disease — Each patient will undergo a blood draw for the analysis of RACH antibodies in serum.
  Also an aliquot of frozen spinal fluid of patient kept in biobank ( spinal fluid taken during a puncture as part of routine care) will be used for the analysis of RACH antibodies.
  Arms: Adults with Alzheimer's disease
Procedure: Adults with Myasthenia — Each patient will undergo a blood draw for the analysis of RACH antibodies in serum.
  Also an aliquot of frozen spinal fluid of patient kept in biobank ( spinal fluid taken during a puncture as part of routine care) will be used for the analysis of RACH antibodies.
  Arms: Adults with Myasthenia
Other: Healhty controls — Frozen spinal fluid of 10 healthy controlled stored in a biobank in Munster, Germanywill be compared to the ones of Adults with Myasthenia and Adults with Alzheimer's disease
  Arms: healthy volonteer

SUMMARY:
The purpose of the study is to evaluate if there is a specific association between the presence of anti Rach antibodies in the CSF and the presence of a cogntive disorder in myasthenic patients. Moreover the investigator wants to study if there is a link between the presence of Anti RACH antibodies in myasthenia and Alzheimers's disease.

For that, the investigator will recruit myasthenic patient with cognitive disorder that has undergo a diagnostic process including lombar punction for memory trouble in Nice memory center as well as Alzheimer's patient having go through the same process.

The study will consist in one additionnal blood draw. Anti RACH antibodies will be analyzed in historical CSF stored in biocollection and serum collected for the study.

LCS of healthy control will also be analyzed.

ELIGIBILITY:
Inclusion criteria

For patient with myasthenia :

1. adult person,
2. Diagnosis of anti-AChR positive autoimmune myasthenia gravis, confirmed by clinical and biological data, and categorized in class I to IV according to the Myasthenia Gravis Foundation of America (MGFA) classification,
3. Mild or major neurocognitive disorder (DSM-5 criterion) having benefited from a diagnosis at the CMRR with CSF biomarker dosage and agreement to bio-collect residual CSF,
4. Agreeing to sign the free and informed consent,
5. Affiliate or beneficiary of a social security system.

For patient with Alzheimer Disease :

1. adult person,
2. Mild or major neurocognitive disorder (DSM-5 criterion) having benefited from a diagnosis at the CMRR with CSF biomarker dosage and agreement to bio-collect residual CSF,
3. Neurocognitive disorder only linked to Alzheimer's disease (IWG-2 criterion): typical or atypical clinical form with biomarkers of Alzheimer's disease in the CSF;
4. Agreeing to sign the free and informed consent,
5. Affiliate or beneficiary of a social security system.

For healty control :

1. absence of memory complaint,
2. absence of neurocognitive disorder,
3. Having agreed to carry out analyzes as part of research, on these CSF samples stored in the biobank of the Institute of Translational Neurology in Münster (Germany)

Exclusion Criteria:

For patient with myasthenia :

1. Person who does not have sufficient command of the French language to understand, read and write, to take neuropsychological tests;
2. Need to use the routine complementary CSF tube to carry out additional diagnostic explorations as part of routine care,
3. Vulnerable people are defined in articles L1121-5 to -8 ( Pregnant women, parturients and breastfeeding mothers, persons deprived of their liberty by a judicial or administrative decision, persons hospitalized without consent under articles L. 3212-1 and L. 3213-1 who do not fall under the provisions of article L. 1121-8, and persons admitted to a health or social establishment for purposes other than research/Adults who are subject to a legal protection measure or who are unable to express their consent.),

For patient with Alzheimer Disease :

1) vulnerable people are defined in articles L1121-5 to -8 ( Pregnant women, parturients and breastfeeding mothers, persons deprived of their liberty by a judicial or administrative decision, persons hospitalized without consent under articles L. 3212-1 and L. 3213-1 who do not fall under the provisions of article L. 1121-8, and persons admitted to a health or social establishment for purposes other than research/Adults who are subject to a legal protection measure or who are unable to express their consent.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The ratio of the number of myasthenic patients with NS-NCD that may be related to myasthenia-related central nervous system damage to the total number of myasthenic patients with CND from all causes combined. | at day 0

SECONDARY OUTCOMES:
Measurement of RACH antibodies in serum | at day 0
  dosage by ELISA method of RACH antibodies
Measurement of RACH antibodies in cerebrospinal liquid | at day 0
  dosage by ELISA method of RACH antibodies

CONTACTS AND LOCATIONS:
Overall Officials: SACCO GUILLAUME, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, Alpes Maritimes, France

IPD SHARING:
Plan to Share IPD: No